CLINICAL TRIAL: NCT06595212
Title: Genetics and Environment iNtersection In the Amyotrophic Lateral Sclerosis - FrontoTemporal Dementia Spectrum: an Italian Twins Cohort studY With a Multi-Omics Approach
Brief Title: Genetics and Environment iNtersection In the ALS-FTD Spectrum: an Italian Twins Cohort studY With a Multi-Omics Approach
Acronym: GENIALITY
Status: Recruiting | Type: Observational
Sponsor: Azienda Ospedaliero-Universitaria di Modena (Other)
Collaborators: A.O.U. Città della Salute e della Scienza - Molinette Hospital (Other); Azienda Ospedaliera Universitaria Policlinico Paolo Giaccone Palermo (Other); University of Modena and Reggio Emilia (Other); Azienda Ospedaliero-Universitaria Careggi (Other)
Responsible Party: Principal Investigator, JESSICA MANDRIOLI, Prof, Azienda Ospedaliero-Universitaria di Modena
Other Study IDs: PNRR-MAD-2022-12375798
Record Dates: First submitted 2024-09-11; First posted 2024-09-19 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2024-09

CONDITIONS: ALS; FTD
Keywords: ALS; FTD; twin; cohort

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Biospecimen Retention: Samples With DNA — blood, CSF (optional), skin, hair, saliva and stool collection
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- affected twins
  Interventions: Other: multiomic profile to assess genetic and environmental risk factiors
- unaffected twins
  Interventions: Other: multiomic profile to assess genetic and environmental risk factiors

INTERVENTIONS:
Other: multiomic profile to assess genetic and environmental risk factiors — Genomic, epigenetic, proteomic, microbiome, immunology, biomarker, metabolite, pesticide, metal, and metalloid investigations will be conducted. The twins will be followed longitudinally from a clinical perspective, with biological sample collections to assess discordance and identify early disease signatures in unaffected individuals.

SUMMARY:
The goal of this study is to learn from discordant twins affected by Amyotrophic Lateral Sclerosis and/or Frontotemporal Dementia the contribution of genetic background versus environmental exposure. The main questions it aims to answer is:

* How far does the genetic background explain the onset of ALS/FTD in discordant twins?
* Which environmental factors and events occurring in post-fetal life influence the onset or progression of this neurodegenerative condition? Participants with ALS and/or FTD with a monozygotic or dizygotic twin willing to contribute to this research will be followed up for two years by specialized Motor Neuron Disorders centers in Italy, donating biological specimen for -omic sciences analysis, and checking out if prodromal signs/symptoms of these two conditions will develop during time.

DETAILED DESCRIPTION:
The main objective of the study is to develop a prospective national twins cohort and virtual biobank collecting demographic, clinical and instrumental data and biological samples of twins with ALS/FTD. Through the definition of a multi-omics profile in ALS twins the study aims to disclose the burden of environmental or genetic risk factors for ALS/FTD and ALS specific biological signatures. Secondary aims include:

* to disclose part of the heritability gap in monozygotic (MZ) discordant twins
* to assess the burden of epigenetic and transcriptomic differences between MZ discordant twins, uncovering which pathways are activated/inactivated in asymptomatic twins and may protect them from the neurodegenerative process
* to evaluate the effects of environment on the risk of developing ALS/FTD (discordant twins) and of developing different phenotypes of ALS (concordant twins). Exposure history will be related to quantification of pesticides, heavy metals and metalloids in biological samples.
* to investigate how lifetime environmental exposures affect microbiota composition and next metabolomics and immune profile
* to correlate biological signatures with clinical features and disease heterogeneity (onset, progression, survival) for discordant twins
* to correlate environmental factors exposure with biological factors as mentioned above (e.g.microbiota, immunological. factors)
* to acquire biological data over time to discriminate between changes related to disease pathogenesis and epiphenomena secondary to the disease advancement.
* to assess neurophysiological, neuropsychological and imaging signatures within the ALS-FTD spectrum of disease across discordant twins, in particular in the asymptomatic twin, in order to disclose potential presymptomatic subclinical traits. In concordant twins, the same extensive batteries will be used to evaluate whether disease progression proceeds at the same pace or affects similar or divergent neuroanatomical substrates.

Study population Being a national ALS-FTD twin cohort study, study population could include all Italian MZ and dizygotic (DZ) twins of whom at least one is affected by ALS or ALS-FTD and possibly their parents for trios studies. ALS/FTD twins will be invited from the referring neurologist to participate in the GENIALITY study and will be sent for screening and baseline visits to the nearest clinical center involved in this study, either Modena, Turin or Palermo.

Twin pairs will undergo a detailed interview, visit, clinical tests including neuropsychological testing (NPS), neuroimaging and neurophysiological studies, extensive environmental and exposure history, and blood, CSF (optional), skin, hair, saliva and stool collection.

ALS patients will be followed up by the centers with visits scheduled every 3-4 months as for clinical practice, while healthy twins will be asked to be followed with neurological evaluations every 6 months up to 24 months of the study duration.

Twins and parents (optional) will be asked to undergo a detailed interview, neurological examination, samples collection (parent-offspring trios studies) including blood sample, saliva and faeces una tantum.

Standard Operating Procedures (SOPs) for sampling, biobanking, clinical, and imaging studies will be shared by all the centers involved in the consortium. SOPs will include requirements for collection, analysis and storage of biological materials and guidelines concerning the shipping of the samples from one center to another, but also guideline concerning the patients' recruitment, informed consent collection, clinical scales, questionnaires administration. Furthermore, a battery of NPS tests will be shared with centers, as well as methods for neurophysiological assessment and requirements for imaging studies (brain MRI and PET).

This project will generate multi-omics parameters and correlated demographic and clinical data in ALS/FTD patients, their co-twins and possibly their parents. Data collected from interviewers, medical record review, and laboratory data, will be recorded in online case report forms.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 yrs
* Presence of MZ or DZ twins in the family both willing to participate in the study and able to provide informed consent
* At least one twin is affected by ALS as defined by Gold Coast Criteria (Shefner et al., 2020) and/or by FTD as defined by Strong and colleagues (Strong et al., 2017)
* Subjects able and willing to comply with study procedures as per protocol
* Subjects able to understand, and capable of providing informed consent at screening visit before any protocol-specific procedures

Exclusion Criteria:

* Unwillingness to perform assessments as stated in the protocol at least during baseline visit for both twins
* Unwillingness to donate biological samples collected at periphery (lumbar puncture excluded) for both twins
* Women who are pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population include all Italian participants with ALS and/or FTD who have a mozygotic or dizygotic twin with (concordant) or without (discordant) the same condition willing to participate in the study. Once the consent is obtained, the twins will be followed up for 24 months in three possible Italian recruiting centres (Modena, Turin, Palermo).
Sampling Method: Non-Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2024-01-29 (Actual); Primary Completion 2026-01-29 (Estimated); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
Environmental/genetic risk/protective factors involved in driving discordance in monozygotic (MZ) twins | 24 months
  Using a multi-omic approach, the investigators will establish a longitudinal cohort of Italian twins affected by ALS/FTD, collecting various samples to compare affected and unaffected twins across multiple biological and phenotypic variables. The aim is to uncover the factors underlying discordance in monozygotic twins, identifying what protects the unaffected twins and what predisposes the affected ones.

CONTACTS AND LOCATIONS:
Locations (3):
- Italy (3):
  - Azienda Ospedaliero-Universitaria di Modena, Modena, Italy
  - Azienda Ospedaliero-Universitaria Policlinico P. Giaccone di Palermo, Palermo, Italy
  - Azienda Ospedaliero-Universitaria Città della Salute e della Scienza di Torino, Torino, Italy

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in any publication, after deidentification (text, tables, figures, and appendices).
Time Frame: Beginning 3 months and ending 5 years following article publication.
Access Criteria: Researchers who provide a methodologically sound proposal.